CLINICAL TRIAL: NCT04506294
Title: Evaluating an eHealth Solution for Screening in Pediatric Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Kentucky (Other); Radiant Creative Group, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 20-017351; R42HD087021 (NIH)
Record Dates: First submitted 2020-07-15; First posted 2020-08-10 (Actual); Results first posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-05

CONDITIONS: Pain; Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Pain; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eScreen Group (Experimental): After randomization at baseline, use eScreen system (child screening component and parent information component) for 6 weeks.
  Interventions: Behavioral: eScreen system
- Usual Care Group (No Intervention): Treatment as usual from baseline. Optional access to the game only (no screening, no parent information component) after completion of T3 assessment (~12 weeks)

INTERVENTIONS:
Behavioral: eScreen system — The eScreen system is composed of a child screening component and a parent information component. The child screening component is delivered via a game-like interface and includes assessment of current pain, PTSS, and functional recovery. Children are asked to play the game at least 3x/week. The parent information component consists of text / email messages sent to parents at least weekly that summarize child ratings and include a link to an online dashboard with additional personalized information for parents.
  Arms: eScreen Group

SUMMARY:
This study will evaluate the predictive validity of a game-based screening system based on child self-report measures.

The core study hypotheses are that (1) in-game assessments will predict problematic recovery (child pain and posttraumatic stress symptoms [PTSS]) and (2) parents in the intervention group will report greater confidence in managing child recovery.

DETAILED DESCRIPTION:
This study will evaluate the predictive validity of a game-based screening system based on child self-report measures.

The core study hypotheses are that (1) in-game assessments will predict problematic recovery (child pain and PTSS) and (2) parents in the intervention group will report greater confidence in managing child recovery.

Study Design:

This study is a randomized controlled trial that will examine validity of eScreen measures (primary aim) and assess the impact of the eScreen system on parent confidence in managing child symptoms and recovery (secondary aim).

At T1, after baseline assessment (questionnaires), children will be randomized to the usual care plus eScreen (eScreen) or usual care alone (Usual Care) groups. In the eScreen group, children will use the game-based screening component and parents the parent information component for 6 weeks. All participants will complete follow-up research assessments by phone, online, or mail at T2 (6 weeks) and T3 (12 weeks). Following their T3 research assessment, child participants in the Usual Care group will have the option to play and provide feedback on the game (with no in-game assessment and no parent information component).

ELIGIBILITY:
Inclusion Criteria:

* Child treated or admitted for injury or illness event that occurred within the past month
* Child has regular access to a compatible (IOS or Android) tablet at home
* Parent has an internet-capable smartphone and can receive text messages on that phone, OR has email account that can receive messages about child status
* Child and parent read or understand English well enough to consent / assent to participation and complete study tasks (e.g., checklists, use of screening system)

Exclusion Criteria:

* Index medical event is due to family violence

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 320 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Kassam-Adams, PhD, Principal Investigator — Center for Injury Research & Prevention, Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - Kentucky Children's Hospital, Lexington, Kentucky
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Will share de-identified individual participant data, at minimum including key variables relevant to describing participants and assessing primary and secondary outcomes.
Supporting Information: Study Protocol
Time Frame: As soon as possible after core study analyses are complete.
Access Criteria: Qualified researchers.

REFERENCES:
- [Background] Kassam-Adams N, Kohser KL, McLaughlin J, Winston F, Marsac ML. Evaluating the Acceptability and Validity of Assessing Pain and Posttraumatic Stress Symptoms in an Adaptable eHealth System for School-Age Children. Clin Pract Pediatr Psychol. 2019 Mar;7(1):9-19. doi: 10.1037/cpp0000261. PMID 31275781

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited 320 participants (160 child/parent dyads) in two large academic medical centers, between March 2021 and April 2022.
Pre-assignment Details: No pre-assignment procedures other than baseline research assessment measures.
Groups:
- eScreen Group: Ill/injured child and one parent are enrolled in the study. After randomization at baseline, child and parent each use the eScreen system (child: game with screening component; parent: information component) for 6 weeks.
  eScreen system: The eScreen system is composed of a child screening component and a parent information component. The child screening component is delivered via a game-like interface and includes assessment of current pain, PTSS, and functional recovery. Children are asked to play the game at least 3x/week. The parent information component consists of text / email messages sent to parents at least weekly that summarize child ratings and include a link to an online dashboard with additional personalized information for parents.
- Usual Care Group: Ill/injured child and one parent are enrolled in the study. Treatment as usual from baseline to 12 weeks. After completion of T3 assessment (~12 weeks), child is given the option of accessing the game only (no screening). No parent information component is provided.
Period: Overall Study
Arm/Group | eScreen Group | Usual Care Group
Started | 214 | 106
Completed | 128 | 84
Not Completed | 86 | 22
Not completed — Lost to Follow-up | 70 | 20
Not completed — Withdrawal by Subject | 16 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | eScreen Group | Usual Care Group | Total
Number analyzed (Participants) | 214 | 106 | 320
Age, Customized [Count of Participants; unit: Participants]
  age 8-17 (child participants) | 107 | 53 | 160
  age 21-30 (parent participants) | 6 | 2 | 8
  age 31-40 (parent participants) | 36 | 23 | 59
  age 41-50 (parent participants) | 45 | 27 | 72
  age 51-60 (parent participants) | 13 | 1 | 14
  age 61-70 (parent participants) | 2 | 0 | 2
  not reported (parent participants) | 5 | 0 | 5
Sex/Gender, Customized [Count of Participants; unit: Participants]
  female - child | 54 | 26 | 80
  female - parent / guardian | 97 | 51 | 148
  male - child | 53 | 26 | 79
  male - parent / guardian | 7 | 2 | 9
  other - child | 0 | 1 | 1
  other - parent / guardian | 0 | 0 | 0
  not reported - child | 0 | 0 | 0
  not reported - parent / guardian | 3 | 0 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black / African American - child | 17 | 13 | 30
  Black / African American - parent | 17 | 12 | 29
  White - child | 70 | 36 | 106
  White - parent / guardian | 73 | 38 | 111
  Asian - child | 3 | 2 | 5
  Asian - parent / guardian | 4 | 1 | 5
  American Indian / Alaska Native - child | 0 | 0 | 0
  American Indian / Alaska Native - parent / guardian | 1 | 0 | 1
  Multiple - child | 9 | 2 | 11
  Multiple - parent / guardian | 3 | 1 | 4
  Other - child | 7 | 0 | 7
  Other - parent / guardian | 6 | 0 | 6
  Not reported - child | 1 | 0 | 1
  Not reported - parent / guardian | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Validity of eScreen Pain Measure as Predictor of Child's Clinically Significant Pain Severity at 6 Weeks
Description: Predictive validity - Area Under the Curve (AUC) in ROC analyses - baseline eScreen Pain Measure score predicting rating >= 6 on 6-week Numerical Rating Scale for Pain Intensity (NRSI)
  Pain at baseline: eScreen Pain Measure score (0-10) On-screen visual analog 'slider' - width & color intensity increase from bottom to top, face of child's avatar (selected by child in eScreen system) anchors lower & upper ends of slider with validated 'no pain' and 'most pain' facial expressions. On-screen instructions: "The bottom of this scale is no pain, and the top is the most pain you can imagine. Slide the marker to show how much pain you feel right now." Child uses touch screen to slide virtual marker, system derives score from 0.000 to 10.000 based on marker location.
  Pain severity at 6 weeks: NRSI >= 6 Verbally-administered, child rates pain by choosing integer from 0 to 10 "where 0 = no pain or hurt and 10 = the most or worst pain/hurt" Rating >=6 validated as clinically significant.
Time Frame: 6 weeks
Population: At 6 weeks no children reported NRSI >=6 (ie clinically significant pain, thus planned analyses could not be conducted.
Groups:
- eScreen Group: After randomization at baseline, child and parent each use the eScreen system (child: game with screening component; parent: information component) for 6 weeks.
  eScreen system: The eScreen system is composed of a child screening component and a parent information component. The child screening component is delivered via a game-like interface and includes assessment of current pain, PTSS, and functional recovery. Children are asked to play the game at least 3x/week. The parent information component consists of text / email messages sent to parents at least weekly that summarize child ratings and include a link to an online dashboard with additional personalized information for parents.
- Usual Care Group: Treatment as usual from baseline to 12 weeks. After completion of T3 assessment (~12 weeks), child is given the option of accessing the game only (no screening). No parent information component is provided.
Arm/Group | eScreen Group | Usual Care Group
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Validity of eScreen Pain Measure as Predictor of Child's Clinically Significant Pain Interference at 6 Weeks
Description: Predictive validity - Area Under the Curve (AUC) in ROC analyses - baseline eScreen Pain Measure score predicting T score >= 65 on 6-wk PROMIS Pain Interference scale Pain at baseline: eScreen Pain Measure score (0-10) On-screen visual analog 'slider' - width & color intensity increase from bottom to top, face of child's avatar (selected by child in eScreen system) anchors lower & upper ends of slider with validated 'no pain' and 'most pain' facial expressions. On-screen instructions: "The bottom of this scale is no pain, and the top is the most pain you can imagine. Slide the marker to show how much pain you feel right now." Child uses touch screen to slide virtual marker, system derives score from 0.000 to 10.000 based on marker location.
  Pain interference at 6 weeks: PROMIS Pediatric Pain Interference T score >=65 Brief questionnaire - Child rates pain interference with daily activities over past 7 days. Ratings lead to normed T scores where >=65 = significant interference.
Time Frame: 6 weeks
Population: This outcome pertains only to children (not parents); only in the eScreen group.
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | eScreen Group | Usual Care Group
Number analyzed (Participants) | 45 | 0
Probability | .756 [.613 to .900] |

3. Primary Outcome: Validity of eScreen Posttraumatic Stress Screen as Predictor of Posttraumatic Stress at 6 Weeks
Description: Predictive validity - Area Under the Curve (AUC) in ROC analyses - baseline eScreen PTSS Screener score predicting whether child meets symptom criteria for posttraumatic stress disorder (PTSD) on 6-wk Child PTSD Symptom Scale for DSM-5 [CPSS-5] eScreen PTSS Screener eScreen uses the Acute Stress Checklist for Children 6-item Short Form (ASC-6) to screen for posttraumatic stress symptoms (PTSS). Scores range from 0 to 12; higher scores indicate greater PTSS severity.
  Child PTSD Symptom Scale for DSM-5 (CPSS-5) 20-item questionnaire assesses DSM-5 criteria for posttraumatic stress disorder (PTSD), scored here to determine whether child meets symptom criteria for PTSD at 6 wks.
Time Frame: 6 weeks
Population: This outcome pertains only to child participants, and only to those in eScreen group.
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | eScreen Group | Usual Care Group
Number analyzed (Participants) | 44 | 0
Probability | .822 [.650 to .994] |

4. Primary Outcome: Validity of eScreen PTSS Screener as Predictor of Impairment From Posttraumatic Stress Symptoms at 6 Weeks
Description: Predictive validity - Area Under the Curve (AUC) in ROC analyses - baseline eScreen PTSS Screener score predicting whether or not child reports impairment from posttraumatic stress symptoms (PTSS) on 6-wk Child PTSD Symptom Scale for DSM-5 [CPSS-5] eScreen PTSS Screener eScreen uses the Acute Stress Checklist for Children 6-item Short Form (ASC-6) to screen for posttraumatic stress symptoms (PTSS). Scores range from 0 to 12; higher scores indicate greater PTSS severity.
  Child PTSD Symptom Scale for DSM-5 (CPSS-5) 7 items in the CPSS questionnaire assess impairment (in social/interpersonal or academic functioning or daily activities) related to posttraumatic stress symptoms. Impairment scored as present if child endorses impairment on any item at 6 wks.
Time Frame: 6 weeks
Population: This outcome pertains only to child participants, and only to those in the eScreen group.
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | eScreen Group | Usual Care Group
Number analyzed (Participants) | 44 | 0
Probability | .691 [.531 to .850] |

5. Secondary Outcome: Impact of eScreen System on Parent Confidence in Managing Child Symptoms and Recovery
Description: Examine difference between eScreen and usual care groups on parents' self-rated confidence (at 6 weeks) related to managing child symptoms and recovery after discharge.
  Parent Confidence Scale - 9 Likert-scale items in which parents rate (from 1 to 5) the extent to which they have felt prepared to manage their ill or injured child's symptoms and recovery after hospital or clinic discharge. Summed total scores range from 5 to 45, higher scores indicate greater confidence.
Time Frame: 6 weeks
Population: This outcome pertains only to parent participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | eScreen Group | Usual Care Group
Number analyzed (Participants) | 68 | 43
score on a scale | 39.6 (5.2) | 38.9 (6.9)
Statistical Analysis 1: Comparison: eScreen Group vs Usual Care Group; Test type: Superiority; p = .536, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Adverse Event definition is same as clinicaltrials.gov definition
Arm/Group | eScreen Group | Usual Care Group
All-Cause Mortality (participants affected / at risk) | 0/214 | 0/106
Serious Adverse Events (participants affected / at risk) | 0/214 | 0/106
Other Adverse Events (participants affected / at risk) | 0/214 | 0/106

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/94/NCT04506294/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/94/NCT04506294/ICF_001.pdf